CLINICAL TRIAL: NCT01971918
Title: Comparative Analysis of Two Therapeutic Strategies: "Early Switch" Versus "Therapeutic Intensification" in Patients With Spondyloarthritis Treated With Anti-tnf Biologics, in Case of Secondary Treatment Failure Suspicion.
Brief Title: Comparative Analysis of Two Therapeutic Strategies in Patients With Spondyloarthritis Treated With Anti-tnf Biologics
Acronym: STRADA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/006/HP
Record Dates: First submitted 2013-10-11; First posted 2013-10-29 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Spondyloarthritis
Keywords: spondyloarthritis; monoclonal antibodies anti-TNF; secondary treatment failure
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early switch (Experimental): * early switch of monoclonal antibodies anti-TNF
  * anti drug antibodies dosage
  Interventions: Biological: anti drug antibodies dosage
- therapeutic intensification (Experimental): * therapeutic intensification of monoclonal antibodies anti-TNF
  * anti drug antibodies dosage
  Interventions: Biological: anti drug antibodies dosage

INTERVENTIONS:
Biological: anti drug antibodies dosage — anti drug antibodies dosage

SUMMARY:
The objective of the study is to evaluate two therapeutic strategies: "early switch" or "therapeutic intensification" in patients with spondyloarthritis in case of secondary treatment failure suspicion to a first monoclonal antibodies anti-TNF definite by increase of ASDAS and positivity to ADAb.

Patients and Methods:

Multicentric randomized prospective study. Duration of inclusion 30 months. Duration of follow-up 24 months. 104 patients with spondyloarthritis treated with infliximab or adalimumab will be included if their ADAb dosage is positive, and they will be randomized (1:1) in two groups : "early switch" where treatment will be change to another anti-TNF, or "therapeutic intensification" where interval between two injections will be shortened. Patients will be evaluated clinically (ASDAS) and biologically (ADAb) at 12 weeks then at 24 weeks. Principal outcome will be the variation of ASDAS between baseline and end of the study. Number of patients to be included has been determined statistically from a preliminary study (power >98% for ASDAS variation of 20% on week 24).

Expected results:

On week 24, we expect a better response and a greater proportion of patients in remission in the "early switch" arm compare to the "therapeutic intensification" arm.

ELIGIBILITY:
Inclusion Criteria:

* Spondyloarthritis positive for the ASAS criteria, treated with a first biologic : infliximab ( 5mg/kg intravenously every 8 weeks) or adalimumab (40mg subcutaneously every 2 weeks)
* Active spondyloarthritis definite by ASDAS-CRP > 2.1 at two successive evaluations while patient was previously responder (ASDAS<2.1 at least once in the 6th months after beginning of treatment)
* Positivity to anti-drug antibodies (ADAb)
* Consent of the patient
* No contra-indication to another anti-tnf biologic
* affiliation to health insurance
* woman of childbearing age must use an appropriate mean of contraception

Exclusion Criteria:

* Pregnant or breastfeeding woman
* contra-indication to anti-tnf biologic
* patient with known hypersensitivity to any of the excipients
* Severe and uncontrolled opportunistic infection , includins septicemia, tuberculosis, abcess and opportunistic infection
* Evolutive infection, including chronic or localised infection
* Patient with moderate to severe heart failure (NYHA class III/IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Variation of ASDAS between inclusion and 24 weeks of treatment | Week 24
  ASDAS will be measured at week 24 and will be compared to day 1

SECONDARY OUTCOMES:
Frequency of patients with ASDAS < 2.1 | Week 24
  Frequency of patients with ASDAS < 2.1 at week 24 ASDAS < 2.1 is considered as remission

OTHER OUTCOMES:
Safety analysis - Occurence of adverse event | Week 24
  safety analysis in each arm at week 24 Safety analysis include occurence of adverse event in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Olivier VITTECOQ, Prof, Principal Investigator — UH Rouen
Locations (7):
- France (7):
  - UH Amiens, Amiens
  - UH Caen, Caen
  - Dieppe Hospital, Dieppe
  - Elbeuf Hospital, Elbeuf
  - UH Lille, Lille
  - Le Havre Hospital, Montivilliers
  - UH Rouen, Rouen